CLINICAL TRIAL: NCT05741281
Title: The Effect of Physical Exercises Program on Social Functioning, Alexithymia and Sense of Coherence Among Patients With Bipolar Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1692022
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Social Functioning, Alexithymia and Sense of Coherence , Bipolar Disorders
MeSH Terms: conditions — Social Adjustment; Affective Symptoms; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): Physical exercises will be carried out for patients in the study group . The physical exercise intervention phase will take three weeks for each patient (three sessions per week for three weeks - Nine sessions for each group). It will be applied for two groups each week for three weeks (one group / day - 3 sessions /week for each group - six days/ week for the two groups).
  Interventions: Behavioral: Physical exercises program
- Control group (Active Comparator): Those in the control group will be left to undergo the usual hospital routine
  Interventions: Behavioral: Physical exercises program

INTERVENTIONS:
Behavioral: Physical exercises program — - Physical exercise program is an innovative exercise program-consisting of three basic parts (warm up - physical fitness - cool down). It was developed previously by the researcher under the supervision of experienced trainer of physical exercise. The session will begin with a 5- to 10-minutes warm-up consisting of stretching and bending movements. This will be followed by physical fitness phase for 30 to 35 minutes which consist of rapid walking accompanied by a variety of arm and leg movements. The session will be ended by a 5- to 10-minutes cool down phase similar to the warm-up. The total time needed for finishing the physical exercise intervention will be approximately 1 hour.

SUMMARY:
The aim of this study is to:

Investigate the effect of applying physical exercises program on social functioning, alexithymia and sense of coherence among patients with bipolar disorders Research Hypotheses

* Clients who participated in physical exercises program will exhibit better social functioning and sense of coherence than the control group.
* Clients who participated in physical exercises program will exhibit less alexithymia than the control group.

DETAILED DESCRIPTION:
* Psychotic male patients' wards will be randomly selected using simple random sampling technique. The first selected ward will be assigned for the first small study group and its control group. The second selected ward will be assigned for the second study and control group and so on. Then the wards will be revisited again in the same order to achieve the required number of subjects.
* Patients' medical charts in the selected wards will be reviewed to identify those who meet the inclusion criteria. From all patients who meet the predetermined inclusion criteria in the selected ward, the patients will be recruited using simple randomization technique.
* A medical checkup will be performed for patients in the study group to exclude any contraindications for carrying out physical exercise.
* The study group (20 patients) will be divided into 4 small groups of 5 patients. Every patient will be interviewed individually to establish rapport and build trustful relationship. Time of each interview will take from 15 to 30 minutes according to patient's familiarity with the researcher, willingness to talk or cooperate and cognitive abilities. By the end of these interviews, the researcher will explain the purpose of the study, and an informed written consent will be obtained from each patient.
* Patients from the study and control groups will be interviewed and observed individually by the researcher to apply the study tools.
* Physical exercises will be carried out for patients in the study group while those in the control group will be left to undergo the usual hospital routine. The physical exercise intervention phase will take three weeks for each patient (three sessions per week for three weeks - Nine sessions for each group). It will be applied for two groups each week for three weeks (one group / day - 3 sessions /week for each group - six days/ week for the two groups).
* Patients' addresses and telephone numbers will be kept in confidential notebook by the researcher after taking their permission to facilitate follow up of patients at the outpatient level to collect data after intervention.
* After termination of the physical exercise program, every patient recruited in both groups will be interviewed immediately using the study tools. In addition, after three months of discharge, patients in both groups will be interviewed and observed at the outpatient level.

ELIGIBILITY:
Inclusion Criteria:

male patients with no co-morbidity, with duration of illness not exceeding 10 years, physically fit to be able to participate in physical exercise (based on physician recommendations), recently admitted (2 - 3 weeks) Exclusion Criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
The Social Functioning Scale (SFS) | 2 weeks
  The SFS is a self-administered questionnaire and consists of 79 items with varying response format (dichotomous questions, three point likert scale, four point likert scale and five point likert scale). These items are classified into seven subscales; withdrawal/social engagement )5 items), interpersonal communication (4 items), independence-performance(13 items), independence-competence (13 items), recreation (15 items), prosocial activities (22 items), and employment/occupation(5 items), in addition to two unscored preliminary questions.
Toronto Alexithymia Scale | 2 weeks
  The Toronto Alexithymia Scale (TAS-20) was developed by (Bagby, Taylor, & Parker, 1994) and it is a 20-items, self-administered questionnaire that measures difficulty in identifying and describing emotions, which is a big part of alexithymia. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. There are 5 items that are negatively keyed (items 4, 5, 10, 18 and 19). The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
The Sense of Coherence | 2 weeks
  The SOC scale was developed by Antonovsky to measure the concept of sense of coherence. The short form of the SOC scale consists of 13 items that comprise three components: comprehensibility (to which 5 items contribute), manageability (4 items), and meaningfulness (4 items). The respondents indicate agreement or disagreement on a 7-category semantic differential scale with two anchoring responses tailored to the content of each item. Five items (1, 2, 3, 5, and 7) are reversed before summing the total score. The total score can range from 13 to 91, and a higher score indicates higher SOC

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No